CLINICAL TRIAL: NCT02789085
Title: ANS Effects of ULF-TENS Stimulation in Patients With and Without TMD
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Davide Pietropaoli, Post Doc, University of L'Aquila
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 45423/30.12.2015
Record Dates: First submitted 2015-12-31; First posted 2016-06-02 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: TEMPOROMANDIBULAR JOINT DISEASES
Keywords: TENS; ULF-TENS; ANS; Dentistry; TMD
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): without tens stimulation
- Test (Experimental): with tens stimulation
  Interventions: Device: ULF TENS stimulation

INTERVENTIONS:
Device: ULF TENS stimulation
  Arms: Test

SUMMARY:
Using computerized pupillometry, previous research established that the autonomic nervous system (ANS) is dysregulated in patients who suffer from temporomandibular disorders (TMDs), suggesting a potential role for ANS dysfunction in pain modulation and the etiology of TMD. However, pain modulation hypotheses in TMD are still lacking.

The periaqueductal gray (PAG) is involved in the descending modulation of defensive behavior and pain through μ, κ, and δ opioid receptors. Transcutaneous electric nerve stimulation (TENS) has been extensively used for pain relief, as low-frequency stimulation is able to activate µ receptors. The aim of the present study is to use ANS polygraph and salivary/serum biomarkers to evaluate the effect of low-frequency TENS stimulation of ANS in TMD patients.

According to the Research Diagnostic Criteria for TMD, people with myogenous TMD and matched-controls will be enrolled. All subjects will be randomly assigned to control group (no tens stimulation) and case group (test stimulation); subsequently, ANS parameters by both biomarkers and ANS polygraph, before, soon after (end of stimulation), and late after (recovery period) sensorial TENS will be collected.

The overall statistics will be performed from all conditions recorded comparing controls vs cases.

The expected results consist in discovering ANS deregulation in TMD with and without TENS stimulation.

DETAILED DESCRIPTION:
Rationale & background information

Transcutaneous Electric Nervous Stimulation (TENS) is extensively used for pain relief. Notably, Ultra Low Frequency TENS (ULF-TENS) has been used both in research and in dentistry as a reliable tool for the diagnosis and treatment of temporomandibular disorders (TMD).

The mechanism of action of TENS has been widely investigated and involves local and systemic effects. In particular, experiments using animal models have shown systemic action trough involvement of the autonomic nervous system (ANS). Endogenous opioid and descending pain modulatory systems are thought to be involved in central activation during TENS stimulation. In particular, pain modulation occurs via endogenous opioids and affects the periaqueductal gray (PAG) and rostral ventromedial medulla (RVM) brain regions. The PAG provides a neuroanatomical and neuro-functional substrate to couple cortical outflow with the adequate autonomic response.

To study ANS activity and responses during conditions of rest and stress, heart rate variability (HRV) and breathing rate (BR) are traditionally used in experiments due to their repeatability and reliability. To study TENS effects on the autonomic nervous system, HRV has been used; however, pupillometry, skin conductance, blood flow and skin temperature, are also reliable indicators that have been used to study ANS.

Data supports the hypothesis that TENS could act on peripheral autonomic effectors via sympathovagal balance and PAG-opioid activity. Moreover, it has been suggested that PAG participates in the medial viscero-motor network that represents the link between emotional and cognitive functions managed by autonomic support. In particular, these neuro-connections is successfully investigated by the use of HRV.

The goal of the present study is to investigate the effects of TENS stimulation on peripheral autonomic behavior during ULF-TENS stimulation. It is hypothesized that TENS reduces the peripheral autonomic indexes.

Study goals and objectives

The goal of the present proposal is to investigate ANS effects of ULF-TENS stimulation in patients with and without TMD conducting an observational RTC. The enrolled subject (with and without TMD) will be randomly assigned to case and control groups. The case group will receive a total of 40 minutes of TENS stimulation, whereas control group will not. ANS of both groups will be investigated by ANS polygraph and by the use of serum/saliva biomarkers such as:

* Total antioxidant capacity (TAC)
* Total pro-oxidant activity (TPA)
* Noradrenaline
* Alpha-amylase.

Methodology • Autonomic data collection

Autonomic data collection will be performed between 9 a.m. and 12 p.m. and with the subjects will stay in a horizontal supine position on a medical bed. Room temperature (21°C), lighting (3200 K; 500 lx according to Uni En 12464), and relative humidity (50%) will be controlled. External and internal noise sources will be excluded. Before recording sessions, patients will be encouraged to urinate and then will be requested to lie on the medical bed for clinical examination with their eyes open for at least 10 minutes to adapt to the room temperature and humidity and also to reduce their anxiety. During this time, the autonomic sensors will be applied and connected to the polygraph. After connection, subjects will be asked to close their eyes and to maintain their position until the end of the recording session. During the entire recording session, data collection will be obtained from each subject using an 8-channel digital polygraph (Procomp Infinity,Thought Technology Ltd, Montreal, Canada).

• HRV collection and analysis

A three electrode (left shoulder, right shoulder and abdomen) electrocardiogram (ECG) will be recorded at a sampling rate of 2048 Hz. Artifacts and heartbeats that will not be generated by sinus node depolarization will be manually edited by an ECG expert who is blinded about the study aims, protocol, and experimental paradigm. Inter beat intervals (IBI) will be automatically calculated from recurrence rate (RR) intervals. Spectral analysis will be carried out using a fast Fourier transform to generate the heart period power spectrum. The heart rate (HR) parameters used were automatically elaborated and included the following: Heart rate (HR); High frequency band (0.15-0.4 Hz, HF n.u.); Low frequency band (0.04-0.15 Hz, LF n.u.); LF/HF ratio, Root Mean Square Standard Deviation (RMSSD); Percentage of the normal sinus-initiates IBI (pNN50); Determinism (DET); and RR.

• Respiratory rate measurement

Respiratory rate measurement will be obtained by a strain gauge worn by the subjects at the tenth rib and will be connected to the polygraph. The rate sampling is 24 Hz. The two highest, subsequent strain values will be used to define the breath frequency rate.

• Surface Electromyography

Surface Electromyography (sEMG) will be recorded through one channel that is sampled at 2048 Hz using a bipolar electrode (Myotronics-Noromed, Inc., Tukwila, WA, USA). The bipolar electrode will be positioned on the skin over the suprahyoid muscle to precisely detect the start and end of TENS and to detect the numbering tasks, thus allowing the correct selection of study epochs.

• TENS procedure

The method for sensory TENS was described previously. Briefly, a J5 Myomonitor TENS Unit device (Myotronics-Noromed, Inc., Tukwila, WA, USA) with disposable electrodes (Myotrode SG Electrodes, Myotronics-Noromed, Inc., Tukwila, WA, USA) will be used. This low-frequency neurostimulator generates a repetitive synchronous and bilateral stimulus delivered at 1.5 s intervals. The stimulus has adjustable amplitude of approximately 0-24 mA, duration of 500 μs, and frequency of 0.66 Hz. Two TENS electrodes will be placed bilaterally over the cutaneous projection of the notch of the fifth pair of cranial nerves, which is located between the coronoid and condylar processes and will be retrieved by manual palpation of the zone anterior to the tragus. Additionally, a third grounding electrode will be placed in the center of the back of the neck. The amplitude of TENS stimulation started at 0 mA, with the stimulator turned on and the rheostat, which controls the amplitude, positioned at 0. The amplitude of stimulation will be progressively increased at a rate of 0.6 mA/s until the patients reported a pricking sensation. The duration of each stimulation will be 40 minutes. Particular attention will be paid to avoid reaching the threshold of motor stimulation; if any movement of the investigated muscles will be observed, the amplitude of stimulation will be immediately reduced.

The same operator (RC) will apply the polygraph and will deliver the TENS, and both will be performed according to the manufacturer's guidelines.

• Recording procedure

Test and control subjects will naive to the trial protocol and will gone identical polygraph and TENS connection procedures. The control group will be connected to the TENS stimulation device in a manner identical to the test subject group; however, in the control group, the TENS stimulation device will remain off.

Study experimental protocol. The study subject will entry the experiment room, and TENS, EEG and EMG electrodes will be placed and will be tested before starting the session. TENS and ANS polygraphs will be tested and setup for the experiment. Then, the patient will be placed on the medical bed with their eyes open to allow for room acclimation. After 10' of room acclimation, the ANS recording session will start. The first 3' will be dedicated to adaptation and software setup; then, ANS data will be recorded for 5' (basal). At this point, the test group (represented by red rectangles) will receive sensorial TENS, whereas the control group (represented by blue rectangles) will not. TENS stimulation will be administered for 40' in total, allowing 1' for adaptation and 39' of useful recording time (T1). The end of TENS stimulation will be followed by 1' of recovery. Finally, the effects of ULF-TENS will be recorded for 5' (recovery). At each phase (Basal, T1, Recovery) serum and saliva will be sampled using a glycemic stick technique and sterile tubes.

* Serum and saliva analysis

All collected samples from saliva and serum will be analyzed simultaneously by the use of specific ELISA kits.

Safety Considerations

All the used electrical devices that will be employed with patients are conformity to ISO 13485 and European guideline in medical safety 93/42/CEE.

All samples will be stored in a refrigerator key locked under the jurisdiction of Prof Annalisa Monaco under the MeSVA unit.

The study database will be designed and created throughout the project year 1. Due to data safety reasons and to comply with the data privacy protection, the personal data of every patient will be pseudonymized. This ensures the strictly split between the personal data and patient-related dataset (trial data).The Remote Data Entry (RDE) system generates automatically a pseudonym for every new patient. The pseudonym will be a combination of six alphanumeric characters. All trial data of the patient will be linked with this pseudonym. Personal data of the patient will not be saved in the trial database at any time. Data required for the analysis will be acquired and transferred electronically to a central database at Dental Unit MeSVA department. This system allows the documentation of study data on electronic case report form (eCRF). Study data will be entered online direct by the sites. The access to the eCRF requires the authentication by the study participants. All access rights (read or enter data) will be defined depending on their function in the study (Principle, clinical investigator, CRA, etc.). At the end of the study the data will be exported from the database.The study data will be prepared for the statistical analysis. This data management process contains the plausibility, consistency, identification of missing data and range checks of the data. Information of missing data will be given to the respective study centre for possible completion or explanation of missing data.

Statistical analysis of outcome measures

Statistical analysis of outcome measures, in dependence of scale level and distribution, according the post-hoc power-calculation will be performed. The statistical power of comparisons between cases and controls are evaluated. Difference in mean will be detected with level of significance 5%. In addition an alpha-adjustment for the entirety of all tests is planned. Also 95% confidence intervals will be calculated. Descriptives for all primary and secondary clinical, demographic and safety parameters will include absolute and relative frequencies for categorial variables and mean, standard deviation, median, and range for quantitative measurements, according the statistical analysis plan (SAP).

Additional subgroup analyses are planned. Controlling for potential confounders will performed by using multiple statistical models adjusting for these variables. The power-calculations and statistical analysis will be performed by Pietropaoli Davide using R and STATA.

Identification of influencing factors and confounders

95% confidence intervals will be calculated. Descriptives for all primary and secondary clinical, demographic and safety parameters will include absolute and relative frequencies for categorial variables and mean, standard deviation, median, and range for quantitative measurements, according the statistical analysis plan (SAP). Additional subgroup analyses are planned. Controlling for potential confounders will performed by using multiple statistical models adjusting for these variables.

ELIGIBILITY:
Inclusion Criteria:

* myogenous TMD;
* pain duration longer than 3 months;
* presence of complete permanent dentition, with the possible exception of the third molars;
* normal occlusion.

Exclusion Criteria:

Patients were excluded from the study if they met one or more of the following criteria:

* presence of systemic or metabolic diseases;
* eye diseases or visual defects;
* history of local or general trauma;
* neurological or psychiatric disorders;
* muscular diseases;
* cervical pain;
* bruxism, as diagnosed by the presence of parafunctional facets and/or anamnesis of parafunctional tooth clenching and/or grinding;
* pregnancy;
* assumed use of anti-inflammatory, analgesic, anti-depressant, opioid, or myorelaxant drugs;
* smoking;
* fixed or removable prostheses;
* fixed restorations that affected the occlusal surfaces;
* and either previous or concurrent orthodontic or orthognathic treatment.

For comparison with previous literature, the diagnosis of myofascial-type TMD was provided after clinical examination by a trained clinician according to group 1a and 1b of the Research Diagnostic Criteria for TMD (RDC/TMD), in a blinded manner

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Between groups difference in ANS activity, expressed as heart rate (HR), as assessed by computed polygraph | Average of 1 year
  HR: heart rate assessed by ANS polygraph (expressed as beats/minute)
Between groups difference in ANS activity, expressed as heart rate variability parameters (HRV, DET, RR), as assessed by computed polygraph | Average of 1 year
  HRV: heart rate variability assessed by ANS polygraph (expressed as pure number); DET: determinism of HRV measurement assessed by KUBIOS software using HRV data (expressed as pure number); RR: recurrence rate assessed by KUBIOS software using HRV data (expressed as pure number).
Between groups difference in ANS activity, expressed as EMG of suprahyoid muscles, as assessed by computed polygraph | Average of 1 year
  EMG: surface electromyography of suprahyoid muscles (expressed in microvolts)
Between groups difference in ANS activity, expressed as breathing rate, as assessed by computed polygraph | Average of 1 year
  breathing rate: assessed by ANS polygraph (expressed as respiratory acts/minute);
Between groups difference in ANS activity, expressed as skin conductance, as assessed by computed polygraph | Average of 1 year
  Skin conductance: assessed by ANS polygraph (expressed in Ohm)
Between groups difference in ANS activity, expressed as skin temperature, as assessed by computed polygraph | Average of 1 year
  Skin temperature: assessed by ANS polygraph (expressed in grades Celsius).

SECONDARY OUTCOMES:
Between groups difference in ANS activity, expressed as total antioxidant capacity (TAC), as assessed by ELISA | Average of 1 year
  TAC: serum total antioxidant capacity assessed by ELISA (expressed as nmol Cu2+ reduced)
Between groups difference in ANS activity, expressed as serum total pro-oxidant activity (TPA) assessed by ELISA | Average of 1 year
  TPA: serum total pro-oxidant activity assessed by ELISA (expressed as nmol Fe2+ oxidized)
Between groups difference in ANS activity, expressed as serum and salivary noradrenaline, as assessed by ELISA | Average of 1 year
  serum and salivary noradrenaline, as assessed by ELISA (expressed in ng/ml)
Between groups difference in ANS activity, expressed as salivary alpha-amylase, assessed by ELISA. | Average of 1 year
  Salivary alpha-amylase assessed by ELISA (expressed in IU/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- Dental Clinic, University of L'Aquila, St. Salvatore Hospital,, L’Aquila, L'Aquila, Italy

REFERENCES:
- [Background] DeSantana JM, Walsh DM, Vance C, Rakel BA, Sluka KA. Effectiveness of transcutaneous electrical nerve stimulation for treatment of hyperalgesia and pain. Curr Rheumatol Rep. 2008 Dec;10(6):492-9. doi: 10.1007/s11926-008-0080-z. PMID 19007541
- [Background] Sluka KA, Walsh D. Transcutaneous electrical nerve stimulation: basic science mechanisms and clinical effectiveness. J Pain. 2003 Apr;4(3):109-21. doi: 10.1054/jpai.2003.434. PMID 14622708
- [Background] Cooper BC; International College of Cranio-Mandibular Orthopedics (ICCMO). Temporomandibular disorders: A position paper of the International College of Cranio-Mandibular Orthopedics (ICCMO). Cranio. 2011 Jul;29(3):237-44. doi: 10.1179/crn.2011.034. PMID 22586834
- [Background] Keay KA, Bandler R. Parallel circuits mediating distinct emotional coping reactions to different types of stress. Neurosci Biobehav Rev. 2001 Dec;25(7-8):669-78. doi: 10.1016/s0149-7634(01)00049-5. PMID 11801292
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Francesco B, Maria Grazia B, Emanuele G, Valentina F, Sara C, Chiara F, Riccardo M, Francesco F. Linear and nonlinear heart rate variability indexes in clinical practice. Comput Math Methods Med. 2012;2012:219080. doi: 10.1155/2012/219080. Epub 2012 Feb 14. PMID 22400047
- [Background] Thayer JF, Lane RD. A model of neurovisceral integration in emotion regulation and dysregulation. J Affect Disord. 2000 Dec;61(3):201-16. doi: 10.1016/s0165-0327(00)00338-4. PMID 11163422
- [Background] Tarvainen MP, Niskanen JP, Lipponen JA, Ranta-Aho PO, Karjalainen PA. Kubios HRV--heart rate variability analysis software. Comput Methods Programs Biomed. 2014;113(1):210-20. doi: 10.1016/j.cmpb.2013.07.024. Epub 2013 Aug 6. PMID 24054542
- [Result] Johnson M, Martinson M. Efficacy of electrical nerve stimulation for chronic musculoskeletal pain: a meta-analysis of randomized controlled trials. Pain. 2007 Jul;130(1-2):157-65. doi: 10.1016/j.pain.2007.02.007. Epub 2007 Mar 23. PMID 17383095
- [Result] Katch EM. Application of transcutaneous electrical nerve stimulation in dentistry. Anesth Prog. 1986 May-Jun;33(3):156-60. PMID 3488697
- [Result] Ainsworth L, Budelier K, Clinesmith M, Fiedler A, Landstrom R, Leeper BJ, Moeller L, Mutch S, O'Dell K, Ross J, Radhakrishnan R, Sluka KA. Transcutaneous electrical nerve stimulation (TENS) reduces chronic hyperalgesia induced by muscle inflammation. Pain. 2006 Jan;120(1-2):182-187. doi: 10.1016/j.pain.2005.10.030. Epub 2005 Dec 19. PMID 16360266
- [Result] DeSantana JM, Da Silva LF, De Resende MA, Sluka KA. Transcutaneous electrical nerve stimulation at both high and low frequencies activates ventrolateral periaqueductal grey to decrease mechanical hyperalgesia in arthritic rats. Neuroscience. 2009 Nov 10;163(4):1233-41. doi: 10.1016/j.neuroscience.2009.06.056. Epub 2009 Jul 2. PMID 19576962
- [Result] Kalra A, Urban MO, Sluka KA. Blockade of opioid receptors in rostral ventral medulla prevents antihyperalgesia produced by transcutaneous electrical nerve stimulation (TENS). J Pharmacol Exp Ther. 2001 Jul;298(1):257-63. PMID 11408550
- [Result] Bandler R, Keay KA, Floyd N, Price J. Central circuits mediating patterned autonomic activity during active vs. passive emotional coping. Brain Res Bull. 2000 Sep 1;53(1):95-104. doi: 10.1016/s0361-9230(00)00313-0. PMID 11033213
- [Result] Lombardi F, Stein PK. Origin of heart rate variability and turbulence: an appraisal of autonomic modulation of cardiovascular function. Front Physiol. 2011 Dec 8;2:95. doi: 10.3389/fphys.2011.00095. eCollection 2011. PMID 22163222
- [Result] Stein C, Dal Lago P, Ferreira JB, Casali KR, Plentz RD. Transcutaneous electrical nerve stimulation at different frequencies on heart rate variability in healthy subjects. Auton Neurosci. 2011 Dec 7;165(2):205-8. doi: 10.1016/j.autneu.2011.07.003. Epub 2011 Aug 9. PMID 21827970
- [Result] Monaco A, Cattaneo R, Mesin L, Ortu E, Giannoni M, Pietropaoli D. Dysregulation of the descending pain system in temporomandibular disorders revealed by low-frequency sensory transcutaneous electrical nerve stimulation: a pupillometric study. PLoS One. 2015 Apr 23;10(4):e0122826. doi: 10.1371/journal.pone.0122826. eCollection 2015. PMID 25905862
- [Result] Monaco A, Cattaneo R, Mesin L, Ciarrocchi I, Sgolastra F, Pietropaoli D. Dysregulation of the autonomous nervous system in patients with temporomandibular disorder: a pupillometric study. PLoS One. 2012;7(9):e45424. doi: 10.1371/journal.pone.0045424. Epub 2012 Sep 18. PMID 23028999
- [Result] Olyaei GR, Talebian S, Hadian MR, Bagheri H, Momadjed F. The effect of transcutaneous electrical nerve stimulation on sympathetic skin response. Electromyogr Clin Neurophysiol. 2004 Jan-Feb;44(1):23-8. PMID 15008021
- [Result] Cramp FL, McCullough GR, Lowe AS, Walsh DM. Transcutaneous electric nerve stimulation: the effect of intensity on local and distal cutaneous blood flow and skin temperature in healthy subjects. Arch Phys Med Rehabil. 2002 Jan;83(1):5-9. doi: 10.1053/apmr.2002.27478. PMID 11782825
- [Result] Xiang XH, Chen YM, Zhang JM, Tian JH, Han JS, Cui CL. Low- and high-frequency transcutaneous electrical acupoint stimulation induces different effects on cerebral mu-opioid receptor availability in rhesus monkeys. J Neurosci Res. 2014 May;92(5):555-63. doi: 10.1002/jnr.23351. Epub 2014 Jan 31. PMID 24482187
- [Result] Sallam H, McNearney TA, Doshi D, Chen JD. Transcutaneous electrical nerve stimulation (TENS) improves upper GI symptoms and balances the sympathovagal activity in scleroderma patients. Dig Dis Sci. 2007 May;52(5):1329-37. doi: 10.1007/s10620-006-9257-3. Epub 2007 Mar 20. PMID 17372833
- [Result] Lane RD, McRae K, Reiman EM, Chen K, Ahern GL, Thayer JF. Neural correlates of heart rate variability during emotion. Neuroimage. 2009 Jan 1;44(1):213-22. doi: 10.1016/j.neuroimage.2008.07.056. Epub 2008 Aug 9. PMID 18778779
- [Result] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Result] Monaco A, Sgolastra F, Pietropaoli D, Giannoni M, Cattaneo R. Comparison between sensory and motor transcutaneous electrical nervous stimulation on electromyographic and kinesiographic activity of patients with temporomandibular disorder: a controlled clinical trial. BMC Musculoskelet Disord. 2013 May 15;14:168. doi: 10.1186/1471-2474-14-168. PMID 23672400
- [Derived] Pietropaoli D, Ortu E, Giannoni M, Cattaneo R, Mummolo A, Monaco A. Alterations in Surface Electromyography Are Associated with Subjective Masticatory Muscle Pain. Pain Res Manag. 2019 Nov 22;2019:6256179. doi: 10.1155/2019/6256179. eCollection 2019. PMID 31885756
- Available data/document: Reference — http://www.psy.unsw.edu.au/research/research-tools/depression-anxiety-stress-scales-dass — UNSW Australia SoP. Depression & Anxiety Stress Scales (DASS): UNSW Australia; 2011